CLINICAL TRIAL: NCT05361681
Title: Assessment of Electromagnetic Interference Between Cardiac Implantable Electronic Devices and High Power Charging Systems for Battery Electric Cars
Brief Title: EMI and CIED: Is High Power Charging of Battery Electric Car Safe?
Acronym: eCarII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GER-EP-024
Record Dates: First submitted 2021-08-31; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-08

CONDITIONS: Pacemaker; ICD

STUDY DESIGN:
Intervention Model Description: Exposure of patients with pacemaker or ICD to the electromagnetic fields of high power charging systems
Masking Description: Assessor is blinded regarding patient and details of intervention (i.e. which charging column and which electric cars were used)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional arm (Experimental): Participants were charging full electric cars, using high power charging systems
  Interventions: Other: Electromagnetic Field Exposure

INTERVENTIONS:
Other: Electromagnetic Field Exposure — All participants were exposed to the electromagnetic field of 4-5 different high power charging systems, charging 4-5 different, commercially available full electric cars

SUMMARY:
It is not known if the use of high power charging systems for electric vehicles may interfere with the functionality of implanted pacemakers and cardioverter-defibrillators.

DETAILED DESCRIPTION:
The use of electric cars for public and private transport is increasing all over the world. Moreover the charging technique is improving and enables very fast charging with the use of high power. It is not known if the use of high volume charging systems interfere with cardiac implantable electronic devices. The study evaluates different types of high volume charging systems connected to different full electric vehicles with regard to electromagnetic interference with implanted pacemakers or cardioverter-defibrillators.

ELIGIBILITY:
Inclusion Criteria:

* implanted cardiac implantable electronic device with regular function

Exclusion Criteria:

* implanted cardiac implantable electronic device with irregular function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Electromagnetic interference | during the intervention, i.e. when participants are exposed to the electromagnetic field of the high power charging column
  Occurence of electromagnetic interference during an exposure time of up to 5 minutes

SECONDARY OUTCOMES:
Electromagnetic fields | during the intervention
  Measuring the electromagnetic fields while super-charging along the charging cable, the column and the car connector

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany